CLINICAL TRIAL: NCT01089946
Title: Cardiovascular Changes and Changes in Tissue Oxygenation During Early Postoperative Mobilization After Primary Total Hip Arthroplasty
Brief Title: Cardiovascular Changes and Changes in Tissue Oxygenation During Early Postoperative Mobilization in Total Hip Arthroplasty (THA) Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Oeivind Jans, M.D, Research Fellow, Rigshospitalet, Denmark
Other Study IDs: RH-4074
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Arthroplasty
Keywords: Mobilization; Hip arthroplasty; cardiovascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the cardiovascular changes during early postoperative mobilization of hip arthroplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Primary THA

Exclusion Criteria:

* Alcoholism
* Known orthostatic hypotension
* Daily use of anxiolytic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary THA.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Orthostatic intolerance | 6 and 24 hours postoperative

SECONDARY OUTCOMES:
Orthostatic hypotension | 6 and 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Oeivind Jans, M.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Hørsholm Hospital, Hørsholm, Denmark

REFERENCES:
- [Result] Jans O, Bundgaard-Nielsen M, Solgaard S, Johansson PI, Kehlet H. Orthostatic intolerance during early mobilization after fast-track hip arthroplasty. Br J Anaesth. 2012 Mar;108(3):436-43. doi: 10.1093/bja/aer403. Epub 2011 Dec 15. PMID 22174345
- [Derived] Jans O, Brinth L, Kehlet H, Mehlsen J. Decreased heart rate variability responses during early postoperative mobilization--an observational study. BMC Anesthesiol. 2015 Aug 22;15:120. doi: 10.1186/s12871-015-0099-4. PMID 26297144